CLINICAL TRIAL: NCT04070664
Title: Evaluation of Thiol/Disulfide Homeostasis and Ischemia Modified Albumin Levels in the Differential Diagnosis of Central and Peripheral Vertigo
Brief Title: Thiol/Disulphide Homeostasis and Albumin in Vertigo
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Alp Şener, Clinical Assistant Professor, Ankara City Hospital Bilkent
Other Study IDs: medybu137
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Vertigo, Peripheral; Vertigo, Central Origin; Oxidative Stress; Diagnosis
Keywords: Vertigo; Central vertigo; Peripheral vertigo; Thiol/disulfide homeostasis; Ischemia modified albumin; Differential diagnosis
MeSH Terms: conditions — Vertigo; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central vertigo: Patients without any pathology on MRI were included in the peripheral vertigo group, and patients whose scans demonstrated acute ischemic infarct in the posterior fossa were included in the central vertigo group.
- Peripheral vertigo: Patients without any pathology on MRI were included in the peripheral vertigo group, and patients whose scans demonstrated acute ischemic infarct in the posterior fossa were included in the central vertigo group.

SUMMARY:
Vertigo is a common complaint in the Emergency Department (ED). The differential diagnosis of central and peripheral vertigo is a difficult issue that directly affects mortality. Magnetic resonance imaging (MRI) is the preferred diagnostic tool, but may not be suitable in all patients due to logistic and economic conditions. In this study, the investigators evaluated the role of thiol/disulfide homeostasis (TDH) parameters and ischemia modified albumin (IMA) levels to assist in the value of being used instead of MRI.

DETAILED DESCRIPTION:
The study was conducted in the ED using a prospective, non-randomized method, and included patients with complaints of acute onset vertigo over 18 years of age and who underwent brain MRI. Pregnant women, smokers, and those with significant neurological signs were excluded. Patients with acute ischemia with MRI were included in the central vertigo group, and patients with normal MRI were included in the peripheral vertigo group. Blood samples for native thiol (NT), total thiol (TT), disulfide, and IMA were collected from all patients at admission. Statistical analyzes were performed with IBM SPSS Statistics for Windows 16.0 Package Program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complaint of vertigo
* Patients over18 years of age

Exclusion Criteria:

* Patients contraindicated for MRI due to metal prosthesis or claustrophobia
* Patients under 18 years of age
* Pregnant patients
* Tobacco users
* Patients exhibiting significant neurological signs or symptoms such as motor or sensory neurologic deficit, speech disorders, unconsciousness, or seizure
* Patients found to have any type of lesion such as a hematoma, mass, cyst, aneurysm, arteriovenous malformation, etc. other than ischemic infarcts on MRI
* Patients with an ischemic lesion other than posterior fossa lesions
* Patients with any type of infection, including upper respiratory tract and ear infections
* Patients previously diagnosed with peripheral vertigo
* Patients where the cause of lightheadedness was blood pressure disorders, cardiac ischemic and arrhythmic disorders, thromboembolic diseases, metabolic disorders, trauma, etc. rather than central and peripheral vertigo.

Ages: 51 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the ED with acute onset vertigo of less than 24 hours and who underwent brain MRI for differential diagnosis of peripheral or central vertigo
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | 6 months
  Thiol/disulphide homeostasis
Ischemic status | 6 months
  Ischemia modified albumin

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, School of Medicine, Department of Emergency Medicine, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing IPD to other researchers.

REFERENCES:
- [Background] Kartal AG, Yilmaz S, Yaka E, Pekdemir M, Sarisoy HT, Cekmen MB, Yuksel M. Diagnostic value of S100B protein in the differential diagnosis of acute vertigo in the emergency department. Acad Emerg Med. 2014 Jul;21(7):736-41. doi: 10.1111/acem.12420. PMID 25125270
- [Background] Bektas H, Vural G, Gumusyayla S, Deniz O, Alisik M, Erel O. Dynamic thiol-disulfide homeostasis in acute ischemic stroke patients. Acta Neurol Belg. 2016 Dec;116(4):489-494. doi: 10.1007/s13760-016-0598-1. Epub 2016 Jan 18. PMID 26782823
- [Background] Sahin E, Deveci I, Dinc ME, Ozker BY, Bicer C, Erel O. Oxidative Status in Patients with Benign Paroxysmal Positional Vertigo. J Int Adv Otol. 2018 Aug;14(2):299-303. doi: 10.5152/iao.2018.4756. PMID 30256204